CLINICAL TRIAL: NCT00881517
Title: Prevention of Human Cytomegalovirus (HCMV) Mother-to-fetus Transmission by Administration of Virus-specific Hyperimmune Globulin to Pregnant Women With Primary HCMV Infection
Brief Title: Efficacy Study of Human Cytomegalovirus (HCMV) Hyperimmune Globulin to Prevent Congenital HCMV Infection
Acronym: CHIP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Maria Grazia Revello, researcher, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FARM7J4HCH
Record Dates: First submitted 2009-04-14; First posted 2009-04-15 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Cytomegalovirus Infection
Keywords: human cytomegalovirus; immune globulin; congenital infection; prevention; pregnancy
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — cytomegalovirus-specific hyperimmune globulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cytotect (Experimental)
  Interventions: Drug: HCMV-specific hyperimmune globulin (Cytotect®)
- placebo (Placebo Comparator)
  Interventions: Drug: Isotonic solution of sodium chloride (placebo)

INTERVENTIONS:
Drug: HCMV-specific hyperimmune globulin (Cytotect®) — 100U (2.0ml)/Kg i.v. every 4 weeks up to 38 weeks' gestation or HCMV-positive amniocentesis or pregnancy termination.
  Other Names: Cytotect®
  Arms: Cytotect
Drug: Isotonic solution of sodium chloride (placebo) — 2.0ml/Kg i.v. every 4 weeks until 38 weeks'gestation or HCMV-positive amniocentesis or pregnancy termination
  Arms: placebo

SUMMARY:
The aim of this trial is to verify, under controlled conditions, the reported efficacy of human cytomegalovirus (HCMV)-specific hyperimmune globulin administration to pregnant women suffering from primary HCMV infection for the prevention of intrauterine HCMV transmission.

DETAILED DESCRIPTION:
HCMV is the leading infectious cause of mental retardation and deafness in infants with congenital HCMV infection. Primary HCMV infections during pregnancy carry the highest risk of fetal infection and disease. No intervention of proven efficacy is available in case of primary HCMV infection in pregnancy. However, a study published in 2005 (Nigro et al., NEJM 353:1350-62, 2005) reported that in pregnant women with primary HCMV infection treated with HCMV-specific hyperimmune globulin (Cytotect®, Biotest) the risk of transmitting the infection to the fetus was reduced from 40% to 16%. Unfortunately, since the study was conducted with inadequate controls, the actual efficacy of hyperimmune globulin could not be properly assessed.

In the present randomized, double-blind, placebo-controlled, multicenter trial pregnant women with ascertained primary HCMV infection at 4-26 weeks of gestation will be randomized to receive Cytotect® or placebo intravenously within 6 weeks after the presumed onset of infection.

Primary efficacy parameter will be the number of HCMV-infected newborns or fetuses.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women (in vitro fertilization permitted)
* >= 18 years of age
* primary HCMV infection at 5-26 weeks' gestation
* <= 6 weeks from presumed onset of infection
* gestational age between 5-32 weeks' gestation
* written informed consent

Exclusion Criteria:

* multiple pregnancy
* history of HIV or HBV or HCV infection
* known immunodeficiency or immunosuppression
* congenital or acquired autoimmune disease
* known intolerance to protein of human origin
* known intolerance to immune globulin
* history of adverse effects to vaccination
* hypersensitivity to human immune globulin (pathological IgG or IgA deficiences)
* renal failure
* serious organic or psychiatric disease
* lack of motivation to participate in the study
* women unable to satisfy study requirements
* women not willing or unable to provide written informed consent
* women not willing to give consent to transmission of anonymised data

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2009-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Evidence of congenital HCMV infection in the fetus/newborn | At amniocentesis and/or within one week after birth

SECONDARY OUTCOMES:
HCMV-specific immune response (humoral and cell-mediated) | 36-48 months
Virological and histological findings in placentas | 36-48 months
Clinical outcome of newborns with congenital HCMV infection | within 2 weeks after birth
Safety of Cytotect in the mother and newborn | within 24 hours after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Maria Grazia Revello, MD, Principal Investigator — SC Ostetricia e Ginecologia, Fondazione IRCCS Policlinico San Matteo, Pavia, Italy
Locations (11):
- Italy (11):
  - Dipartimento di Ostetricia e Ginecologia, Ospedali Riuniti, Bergamo
  - Medicina dell'Età Prenatale, Ospedale Policlinico S.Orsola, Bologna
  - Medicina Materno-Fetale, Spedali Civili, Brescia
  - UOC Malattie Infettive, IRCCS Istituto G.Gaslini, Genova
  - Dipartimento per la salute della donna, del bambino e del neonato. Ospedale Maggiore Policlinico Mangiagalli e Regina Elena, Milan
  - Ostetricia e Ginecologia, Ospedale V.Buzzi, Milan
  - Struttura Semplice di Ostetricia, Ospedale Niguarda Cà Granda, Milan
  - Clinica Ostetrica e Ginecologica, Ospedale S. Gerardo, Monza
  - Ostetricia e Ginecologia, Fondazione IRCCS Policlinico San Matteo, Pavia
  - SCDU Ostetricia e Ginecologia a indirizzo materno fetale, Dipartimento di Discipline Ginecologiche e Ostetriche, Università di Torino, Torino
  - Dipartimento di Ostetricia e Ginecologia, IRCCS Burlo Garofolo, Trieste

REFERENCES:
- [Derived] Revello MG, Lazzarotto T, Guerra B, Spinillo A, Ferrazzi E, Kustermann A, Guaschino S, Vergani P, Todros T, Frusca T, Arossa A, Furione M, Rognoni V, Rizzo N, Gabrielli L, Klersy C, Gerna G; CHIP Study Group. A randomized trial of hyperimmune globulin to prevent congenital cytomegalovirus. N Engl J Med. 2014 Apr 3;370(14):1316-26. doi: 10.1056/NEJMoa1310214. PMID 24693891